CLINICAL TRIAL: NCT05231239
Title: Transcranial Direct Current Stimulation to Reduce Chronic Pelvic Pain in Endometriosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Magdalena S. Prüß née Volz, Principal Investigator ; PD Dr. med., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EA1/174/19
Record Dates: First submitted 2022-01-28; First posted 2022-02-09 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS (Active Comparator): tDCS will be applied for 20 min with 2 mA
  Interventions: Device: tDCS : Transcranial direct current stimulation
- Placebo tDCS (Placebo Comparator): tDCS will be applied for only 20 sec, monatge will be left on the head for 20 min
  Interventions: Device: tDCS : Transcranial direct current stimulation

INTERVENTIONS:
Device: tDCS : Transcranial direct current stimulation — Transcranial direct current stimulation

SUMMARY:
In the study it will be tested whether transcranial direct current stimulation can reduce the perception of pelvic pain in patients with endometriosis.

Hypothesis: Transcranial direct current stimulation can reduce the perception of pelvic pain in patients with patients with endometriosis.

ELIGIBILITY:
Inclusion Criteria:

Endometriosis Chronic pain (more than 3 months) Pain (VAS > 3/10)

Exclusion Criteria:

- Contraindication to transcranial direct current stimulation Pregnancy Sever internal or psychiatric condition

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Pelvic pain via pressure pain threshold | 4 weeks
  pressure pain threshold

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena S Prüß, MD, Principal Investigator — Charite University Medicine Berlin, Germany, 12200
Locations (1):
- Charite University Medicine, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mechsner S, Grunert J, Wiese JJ, Vormbaumen J, Sehouli J, Siegmund B, Neeb L, Pruss MS. Transcranial direct current stimulation to reduce chronic pelvic pain in endometriosis: phase II randomized controlled clinical trial. Pain Med. 2023 Jul 5;24(7):809-817. doi: 10.1093/pm/pnad031. PMID 36882181